CLINICAL TRIAL: NCT04113577
Title: COgilus Remediation in Alzheimer Patients
Brief Title: COgilus Remediation in Alzheimer Patients (CORA)
Acronym: CORA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2019/39
Record Dates: First submitted 2019-10-01; First posted 2019-10-02 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Patient Satisfaction; Neurocognitive Disorders
Keywords: old people; elderly; minor neurocognitive disorder; major neurocognitive disorder; neurocognitive disorder; mild cogntitive impairment; MCI; alzheimer disease; app; usability; ergonomic; satisfaction
MeSH Terms: conditions — Patient Satisfaction; Neurocognitive Disorders; Alzheimer Disease; Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- geriatric inpatients with neurocognitive disorder: usability assessment after 30 minutes to test the app
  Interventions: Other: usability survey
- unformal cargivers: usability assessment after 30 minutes to test the app with their relatives
  Interventions: Other: usability survey
- health professionals: usablity assessment after the enrollement of all patients and unformal caregivers
  Interventions: Other: usability survey

INTERVENTIONS:
Other: usability survey — usability survey composed of subpart: System Usability Scale, questions about global ergonomics of the app, questions about eronomics of the exerecices, question about global satisfaction.

SUMMARY:
This study evaluates the usability of a new tablet PC application to stimulate cognitive functions. Patients hospitalized in a geriatric ward (day or complete hospitalisation) but also their informal and professional caregivers will assess the usability of the application using a structured survey.

DETAILED DESCRIPTION:
Attention span is one of the most frequently and early impaired cognitive functions during aging, especially in neurocognitive disorders such as Alzheimer's disease. Decline of attention span can lead to a cognitive complaint by the patient or his or her relatives, even in the prodromal phase of the disease (DSM V: minor neurocognitive disorder). The current challenge is to develop strategies to prevent the cognitive decline in patients with minor neurocognitive disorder or major cognitive disorder with slight impairment, and thus to limit cognitive decline. However, to date, no strategy has shown clear effectiveness in preventing cognitive decline in patients with neurocognitive disorder.

Interestingly, the integration of perceptual skills are modified in patients with neurocognitive disorders, and in particular visuomotor skills (from early stages). Measurements of evoked potientials during visual stimulation in patients with minor neurocognitive disorder have shown a preservation of sensory responses but a decrease in cognitive responses. Based on this observation, a US team had recently tested the effectiveness of computer-based visual cognitive exercises performed regularly for 8 weeks in patients free of major neurocognitive disorder. They had reported an improvement in information processing speed and walking performance. These results suggest that regular cognitive stimulation exercises using tablet PC visual exercices could improve attention span and in particular the information processing speed in patient with minor or early major neurocognitive disorder.

In particular, Cogilus, a cross-platform tablet PC application (Android, iOS, Microsoft) has recently been developed for this purpose. The Cogilus project, is designed for health professionals who support patients with neurological syndromes including cognitive or attentional dysfunctions. The application is also open to carers and family members, who will be able to support the patient in using the application (based on the exercices proposed by professionals).

The finale objective of the Cogilus project is to assess the impact of the regular use of Cogilus on patient with minor or early major neurocognitive disorder. Considering the specific needs in usability for this population, the first step to devoloppe such technology is to assess the usability of the application in patients but also in unformal and professional cargivers.

ELIGIBILITY:
Inclusion Criteria:

* no opposition to be part of the study
* patients:
* over 65 years old
* to be hospitalised in geriatric medicine department of Angers University Hospital
* mild cognitive impairment (winblad criterion) or minor neurocognitive disorder du to alzheimer disease or early major neurocognitive disorder du to alzheimer disease (DSM V and NINCDS-ADRDA criterion)
* unformal cargivers and health profesionnals:
* over 18 years old

Exclusion Criteria:

* depression (geriatric depression scale 15 items: over 10/15)
* delirum (assessed with the confusion assessment methode)
* to be under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients are recruited during their complet or day hospitalisation in geriatric medicine.
  Relatives / unformal caregivers are recruited during the hospitalisation of patients in geriatric medicine. Professionnal caregivers are recruited in the acute care geriatric unit or in the day hospitalisation geriatric unit.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-10-30 (Estimated); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
Usability regarding the Cogilus app | after 30 minutes of test of the app
  Average of the usability scores. Usability score is calculated using the responses to the validated System Usability Scale (SUS). SUS is composed of 10 questions. Each response is ranking from 0 to 5. The total score ranges between 0 and 100. It is calculted considering the sum of the result on each question multiplicated by 2. An average score equal or over 70/100 will be considered as satisfying.

SECONDARY OUTCOMES:
Satisfaction regarding the Cogilus app | after 30 minutes of test of the app
  Average recommendation score. Satisfaction score is calculated using the responses to the recommendation scale. This scale is a ten point's scale from 0 (I don't recommend at all) to 10 (I fully recommend). An average score greater than 5/10 would be acceptable, a score greater than or equal to 7/10 would be satisfactory.
Global ergonomics regarding the Cogilus app | after 30 minutes of test of the app
  Average ergonomics score: The ergonomics score is a composite score based on the average of the answers to four ergonomics questions on a four-level Likert scale. The Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree). The average score is reported on ten. An average score greater than 5/10 would be acceptable, a score greater than or equal to 7/10 would be satisfactory.
Ergonomics regarding the exercices proposed in the Cogilus app | after 30 minutes of test of the app
  Average ergonomics score: The ergonomics score is a composite score based on the average of the answers to four ergonomics questions on a four-level Likert scale. The Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree). The average score is reported on ten. An average score greater than 5/10 would be acceptable, a score greater than or equal to 7/10 would be satisfactory.

CONTACTS AND LOCATIONS:
Overall Officials: Cedric ANNWEILER, MD, PhD, Principal Investigator — Angers University Hospital
Locations (1):
- Angers University Hospital, Angers, France